CLINICAL TRIAL: NCT03411369
Title: A Randomized, Double Blind, Placebo Controlled Study To Evaluate The Effectiveness Of A Food Supplement Containing Creatine And D-Ribose In Increasing Stress Tolerance In Patients With Ischemic Heart Disease
Brief Title: Creatine, D-Ribose, B1 Vitamin, and B6 Vitamin in Ischemic Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 23473
Record Dates: First submitted 2018-01-10; First posted 2018-01-26 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Ischemic Heart Disease
Keywords: Creatine, ribose, ischemic heart disease.
MeSH Terms: conditions — Myocardial Ischemia | interventions — Creatine; Ribose; Thiamine; Vitamin B 6

STUDY DESIGN:
Intervention Model Description: Two groups, one receiving treatment (Creatine, D-Ribose, B1 Vitamin, and B6 vitamin), and one receiving placebo.
Who Masked: Participant, Investigator
Masking Description: Double blind study design. The dietary supplement of Creatine, D-Ribose, B1 Vitamin, and B6 vitamin will come in the form of water-soluble powder in sachets of 4 grams. Each sachet contains 1 gram of Creatine, 2.5 grams of D-Ribose, 0.33 mg of B1 vitamin and 0.42 mg of B6 vitamin. The same administration will come for placebo group with the inert product sachets consisting of starch powder.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creatine, D-Ribose, B1 Vitamin, and B6 vitamin (Experimental): Water-soluble powder in sachets of 4 grams. Each sachet contains 1 gram of Creatine, 2.5 grams of D-Ribose, 0.33 mg of B1 vitamin and 0.42 mg of B6 vitamin.
  Interventions: Dietary Supplement: Creatine, D-Ribose, B1 Vitamin, and B6 vitamin
- Placebo (Placebo Comparator): Water-soluble powder in sachets of 4 grams containing inert product consisting of starch powder.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine, D-Ribose, B1 Vitamin, and B6 vitamin — The treatment will consist of taking 2 sachets / day for the first two weeks, and then continuing with 1 sachet/day for the next month.
  Other Names: Crebox
  Arms: Creatine, D-Ribose, B1 Vitamin, and B6 vitamin
Other: Placebo — Water-soluble powder in sachets of 4 grams containing inert product consisting of starch powder.
  Arms: Placebo

SUMMARY:
Recently, researchers have paid attention to the development of new products such as supplements food and nutraceuticals for identify and develop integrative therapies to be used in cardiovascular disease. As suggested by literature, some nutritional components (creatine, ribose) can enhance the fundamental energy levels for the functioning of the heart muscle and can enhance the body's antioxidant capacity through the reduction in free radicals activity, one of the main pathogenic mechanisms of these diseases. In this context, the investigators have developed a research with the principal purpose to establish whether a supplement of creatine and ribose can improve the total work capacity during exercise in a population of patients with known ischemic heart disease.

DETAILED DESCRIPTION:
The investigators will enroll patients with previous acute coronary syndrome treated for at least 30 days by hospital discharge. The treatment regimen of all patients will be optimized in accordance with European Society of Cardiology guidelines. Standardized pharmacological treatment during cardiac rehabilitation period will include administration of angiotensin converting enzyme inhibition (ACE), beta-blockers and antiplatelet blockers. Furthermore, in order to keep patients free from angina symptoms, in some cases calcium channel blockers and/or nitrates will be used. The investigators will randomize participants into two groups, one receiving treatment Creatine, D-Ribose, B1 Vitamin, and B6 vitamin, and one receiving placebo in a double blind study design, for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* All patients presented acute coronary syndrome treated with at least 30 days by hospital discharge

Exclusion Criteria:

* oncological diseases
* stable atrial fibrillation
* stent in the common core
* patients who are not able to perform physical activities
* patients with documented sustained ventricular arrhythmias
* pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Blood glucose | Change from Baseline at 6 months
  mg/dl
Total cholesterol | Change from Baseline at 6 months
  mg/dl
LDL-cholesterol | Change from Baseline at 6 months
  mg/dl
HDL-cholesterol | Change from Baseline at 6 months
  mg/dl
Triglycerides | Change from Baseline at 6 months
  mg/dl
Creatinine | Change from Baseline at 6 months
  mg/dl
Alanine transaminase | Change from Baseline at 6 months
  UI/l
Water composition | Change from Baseline at 6 months
  Percentage
Fat mass | Change from Baseline at 6 months
  Percentage
Free fat mass | Change from Baseline at 6 months
  Percentage
Chronotropic index | Change from Baseline at 6 months
  bpm
Cardiac double product at the peak of the load | Change from Baseline at 6 months
  It will be calculated by multiplying systolic blood pressure and heart rate

SECONDARY OUTCOMES:
Body Mass Index | Change from Baseline at 6 months
  Kg/m2
Systolic Blood Pressure | Change from Baseline at 6 months
  mmHg
Heart Rate | Change from Baseline at 6 months
  bpm

IPD SHARING:
Plan to Share IPD: No